CLINICAL TRIAL: NCT04922541
Title: Multi-center Observational Study on the Progression of Atherosclerotic Plaques in Anti-PD-1 mAb Treated Tumor Patients by Artery Ultrasound Follow-up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Cancer Hospital (Other); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); Sun Yat-sen University (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Ningbo No.2 Hospital (Other); Huizhou Municipal Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: #2019-221
Record Dates: First submitted 2021-06-05; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Plaque, Atherosclerotic; Programmed Cell Death Protein 1 Inhibitor
Keywords: atherosclerotic plaque; PD-1 inhibitor; artery ultrasound
MeSH Terms: conditions — Plaque, Atherosclerotic | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: PD-1 inhibitor — dosage form: intravenous injection; frequency: 2-3 weeks; duration: at least 3 months

SUMMARY:
Multi-center Observational Study on the Progression of Atherosclerotic Plaques in Anti-PD-1 mAb Treated Tumor Patients by Artery Ultrasound Follow-up

DETAILED DESCRIPTION:
This is a self-control, multi-center observational study. This study aims to evaluate the effectiveness of anti-PD-1 mAbs on atherosclerotic plaques in those anti-PD-1 mAbs treated patients. The method for quantification and evaluation of atherosclerotic plaques are based on the calculation of the plaque area of atherosclerotic plaques on the long axis direction of artery on the ultrasound images. By comparing the plaque areas at the same location of artery in each patient before and after anti-PD-1 mAbs treatments, to assess the progression of atherosclerotic plaques response to anti-PD-1 mAbs.

ELIGIBILITY:
Inclusion Criteria:

1. The age is 18-90 years old (including 18 and 90 years old);
2. The subjects knew about the experiment and signed the informed consent voluntarily;
3. The subjects complicated with tumor diseases and atherosclerotic plaques;
4. The subjects received regular PD-1 inhibitor treatment;
5. The subjects had ultrasound images of atherosclerotic plaques before- and after- or during PD-1 blockade treatment at the two different timepoints;
6. The subjects received regular treatments of PD-1 inhibitor during the two timepoints of artery ultrasound examinations;
7. The subjects who had ultrasound images before the initiation of first-dose PD-1 inhibitor, the interval between these two timepoints should be restricted within 1 month;
8. The subjects who had ultrasound images after 3 months of PD-1 inhibitor treatment.

Exclusion Criteria:

1. Subjects stop receiving PD-1 inhibitor treatments during follow-up;
2. Subjects are reluctant to continue to be involved in this study; Known pregnant and lactating women;
3. Plaque areas can not be calculated because of the quality of ultrasound image;
4. Other situations that the researchers judged were not suitable for inclusion.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population are the PD-1 inhibitor treated tumor patients from selected multi-center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Sizes of plaque areas at the same locations on artery ultrasound | at least of 3 months after the first dosage of anti-PD-1 mAbs
  Comparison of the sizes of plaque areas at the same locations on artery ultrasound before and after anti-PD-1 mAbs treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine at Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided